CLINICAL TRIAL: NCT05287113
Title: A Randomized, Double-Blind, Multicenter, Phase 2 Study of Retifanlimab in Combination With INCAGN02385 (Anti-LAG-3) and INCAGN02390 (Anti-TIM-3) as First-Line Treatment in Participants With PD-L1-Positive (CPS ≥ 1) Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of Retinfanlimab in Combination With INCAGN02385 and INCAGN02390 as First-Line Treatment in Participants With PD-L1-Positive (CPS ≥ 1) Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCAGN 2385-203; 2023-504270-38-00 (Registry Identifier: EU CT Number); 2021-005775-39 (EudraCT Number)
Expanded Access: NCT06910137 (Available)
Record Dates: First submitted 2022-03-11; First posted 2022-03-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer
Keywords: squamous cell carcinoma of the head and neck (SCCHN); INCAGN02385; INCAGN02390; Retifanlimab; IgG1κ monoclonal antibody; LAG-3; TIM-3; PD-1; PD-L1
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to 1 of 3 treatment groups.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Group 1: Retifanlimab Monotherapy (Experimental): Retifanlimab will be administered intravenously every 4 weeks. Placebos for INCAGN02385 and INCAGN02390 will be administered intravenously every 2 weeks.
  Interventions: Drug: Retifanlimab; Drug: Placebo
- Treatment Group 2: Retifanlimab + INCAGN02385 (Experimental): Retifanlimab will be administered intravenously every 4 weeks. INCAGN02385 and Placebo for INCAGN02390 will be administered intravenously every 2 weeks.
  Interventions: Drug: Retifanlimab; Drug: INCAGN02385; Drug: Placebo
- Treatment Group 3: Retifanlimab + INCAGN02385 + INCAGN02390 (Experimental): Retifanlimab plus INCAGN02385 and INCAGN02390 will be administered intravenously. Retifanlimab will be administered intravenously every 4 weeks. INCAGN02385 and INCAGN02390 will be administered every 2 weeks.
  Interventions: Drug: Retifanlimab; Drug: INCAGN02385; Drug: INCAGN02390

INTERVENTIONS:
Drug: Retifanlimab — Retifanlimab 500mg will be administered intravenously every 4 weeks.
Drug: INCAGN02385 — INCAGN02385 350mg will be administered intravenously every 2 weeks.
  Arms: Treatment Group 2: Retifanlimab + INCAGN02385; Treatment Group 3: Retifanlimab + INCAGN02385 + INCAGN02390
Drug: INCAGN02390 — INCAGN02390 400 mg will be administered intravenously every 2 weeks.
  Arms: Treatment Group 3: Retifanlimab + INCAGN02385 + INCAGN02390
Drug: Placebo — Placebo will be administered intravenously.
  Arms: Treatment Group 1: Retifanlimab Monotherapy; Treatment Group 2: Retifanlimab + INCAGN02385

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the combination of retifanlimab plus INCAGN02385 and retifanlimab plus INCAGN02385 and INCAGN02390 compared with retifanlimab alone as first-line treatment in PD-L1-positive and systemic therapy-naive recurrent/metastatic (R/M) squamous cell carcinoma of the head and neck (SCCHN).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed R/M SCCHN that is not amenable to therapy with curative intent. Participants who refuse potentially curative salvage surgery for recurrent disease are ineligible.
* Eligible primary tumor locations are oropharynx, oral cavity, hypopharynx, and larynx.
* Participants must not have received prior systemic therapy for R/M SCCHN.
* PD-L1 positive tumor status defined by CPS ≥ 1% per central laboratory determination.
* For participants with primary oropharyngeal tumors, documentation of HPV p16 status based on local institutional standard is required. HPV p16 status is not required for other eligible SCCHN primary tumor sites.
* Participant must have at least 1 measurable tumor lesion per RECIST v1.1.
* Availability of archival tissue for biomarker analysis from a core or excisional biopsy or willingness to undergo a fresh biopsy.
* ECOG performance status of 0 or 1.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Progressive or recurrent disease within 6 months of the last dose of systemic treatment for locally advanced SCCHN. Prior PD-(L)1, LAG-3, or TIM-3 directed therapy, or any other checkpoint inhibitor therapy, for SCCHN or any other malignancy.
* Treatment with anticancer therapies or participation in another interventional clinical study within 21 days before the first administration of study treatment.
* Presence of tumors that invade major blood vessels, as shown unequivocally by imaging, and with active bleeding.
* Participants with primary tumors of the nasopharynx, sinonasal cavity, or salivary and are excluded.
* Less than 3-month life expectancy.
* Participant has not recovered to ≤ Grade 1 or baseline from residual toxicities of prior therapy.
* Participant has not recovered adequately from toxicities and/or complications from surgical intervention before starting study treatment.
* Palliative radiation therapy administered within 1 week before the first dose of study treatment or radiation therapy in the thoracic region that is > 30 Gy within 6 months before the first dose of study treatment.
* Known active CNS metastases and/or carcinomatous meningitis. Participants will be excluded if it has been < 4 weeks since radiation therapy was delivered to the CNS.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 24 months
  Defined as the interval between the date of first dose of study treatment and the earliest date of disease progression, based on investigator assessment per RECIST v1.1, or death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  Defined as having a Complete Response (CR) or Partial Response (PR), determined based on investigator assessment per RECIST v1.1.
Duration of Response (DOR) | Up to 24 months
  Defined as the time from earliest date of disease response (CR or PR) until earliest date of disease progression, based on investigator assessment per RECIST v1.1, or death from any cause if occurring sooner than progression.
Disease Control Rate (DCR) | Up to 24 months
  Defined as having CR, PR, or SD (≥ 6 months) as best response, based on investigator assessment per RECIST v1.1.
Overall Survival (OS) | Up to 36 months
  Defined as the interval between the date of the date of first dose of study treatment until death due to any cause.
Participants with treatment-emergent adverse events (TEAE) | Up to 24 months
  TEAE is defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug

CONTACTS AND LOCATIONS:
Locations (91):
- United States (24):
  - Mayo Clinic Rochester, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - City of Hope Orange County, Irvine, California
  - University of California San Diego Medical Center, Moores Cancer Center, La Jolla, California
  - City of Hope-Antelope Valley, Lancaster, California
  - Innovative Clinical Research Institute, Long Beach, California
  - City of Hope National Medical Center, Long Beach, California
  - University of California San Francisco Comprehensive Cancer Center, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Blessed Health Care, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Illinois At Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Hospital Authority, Kansas City, Kansas
  - University of Maryland-Greenebaum Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Hospital, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Huntsman Cancer Institute At University of Utah, Salt Lake City, Utah
  - University of Virginia - Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
- Belgium (3):
  - Grand Hospital de Charleroi, Charleroi
  - Jessa Ziekenhuis, Hasselt
  - Gza Sint Augustinus, Wilrijk
- Canada (3):
  - McGill University Health Centre/Glen Site/Cedars Cancer Centre, Montreal, Quebec
  - Chum Hospital Notre Dame, Montreal, Quebec
  - McGill University Jewish General Hospital, Montreal, Quebec
- France (5):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Institut Curie, Paris
  - Centre Eugene Marquis, Rennes
  - Centre de Lutte Contre Le Cancer - Institut de Cancerologie de L'Ouest - Rene Gauducheau, Saint-Herblain
  - Icans - Institut de Cancerologie Strasbourg Europe, Strasbourg
- Georgia (4):
  - Jsc Evex Hospitals, K'ut'aisi
  - New Hospitals, Tbilisi
  - Jsc Evex Corporation-Caraps Medline, Tbilisi
  - Ltd Cancer Research Centre, Tbilisi
- Germany (4):
  - University of Cologne, Cologne
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
- Greece (4):
  - University Hospital of West Attica - Attikon, Chaïdári
  - Theagenio Anticancer Hospital, Thessaloniki
  - Bioclinic Thessaloniki (Galinos Clinic), Thessaloniki
  - Saint Lukas Clinic, Thessaloniki
- Italy (7):
  - Fondazione Del Piemonte Per L Oncologia Ircc Candiolo, Candiolo
  - Fondazione Irccs Istituto Nazionale Del Tumori Di Milano, Milan
  - European Institute of Oncology, Milan
  - Istituto Nazionale Tumori Irccs Fondazione Pascale, Naples
  - Iov - Istituto Oncologico Veneto Irccs, Padua
  - Fondazione Irccs Policlinico San Matteo, Pavia
  - Ausl-Irccs Di Reggio Emilia, Reggio Emilia
- Netherlands (2):
  - The Dutch Cancer Institue, Amsterdam
  - Leids Universitair Medisch Centrum (Lumc) (Leiden University Medical Center), Leiden
- Poland (6):
  - Centrum Onkologii Im. Prof. Franciszka Lukaszczyka, Bydgoszcz
  - Przychodnia Lekarska Komed Roman Karaszewski, Konin
  - Centrum Onkologii Ziemi Lubelskiej Im. SW. Jana Z Dukli, Lublin
  - Poznan University of Medical Sciences, Poznan
  - Nzoz Provita Prolife Centrum Medyczne, Tomaszów Mazowiecki
  - Centrum Onkologii - Instytut Im. Marii Sklodowskiej - Curie, Warsaw
- Portugal (6):
  - Hospital de Braga, Braga
  - Centro Hospitalar Universitario Algarve, Faro
  - Centro Hospitalar de Lisboa Norte E.P.E. - Hospital de Santa Maria, Lisbon
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil E.P.E., Porto
  - Centro Hospitalar de Sao Joao Alameda, Porto
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, Epe-Unidade L, Vila Nova de Gaia
- South Korea (8):
  - Pusan National University Yangsan Hospital, Busan
  - Chonnam National University Hwasun Hospital, Gwangju
  - Cha Bundang Medical Center, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Kunkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (10):
  - Catalans Institute of Oncology Barcelona, Barcelona
  - Ico Girona Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Fundacion Jimenez Diaz University Hospital, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario Quironsalud Madrid, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari I Politecnic La Fe, Valencia
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation. Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Institutional Review Board Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: Study of Retinfanlimab in Combination With INCAGN02385 and INCAGN02390 as First-Line Treatment in Participants With PD-L1-Positive (CPS ≥ 1) Recurrent/ Metastatic Squamous Cell Carcinoma of the Head and Neck — https://incyteclinicaltrials.com/studies/incagn-2385-203